CLINICAL TRIAL: NCT04394234
Title: Comparative Risk Assessment of Severe Uterine Bleeding Following Exposure to Direct Oral Anticoagulants: A Network Study Across 4 US Observational Databases
Brief Title: A Study of Severe Uterine Bleeding Following Exposure to Direct Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108824; PCSCVM002566 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Uterine Hemorrhage
MeSH Terms: conditions — Uterine Hemorrhage | interventions — N(4)-oleylcytosine arabinoside; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Group: Participants data who are new users of rivaroxaban, apixaban and dabigatran with prior Non-valvular atrial fibrillation/Venous thromboembolism/Total hip replacement (NVAF/VTE/THR) or Total knee replacement (TKR) in a nationally representative population of insured participants in the United States (US) will be compared pairwise.
  Interventions: Drug: Direct oral anticoagulant (DOACs)
- Comparator Group: Participants data who are new users of warfarin, apixaban, and dabigatran with prior NVAF/VTE/THR or TKR in a nationally representative population of insured participants in the US will be compared pairwise.
  Interventions: Drug: Direct oral anticoagulant (DOACs); Drug: Warfarin

INTERVENTIONS:
Drug: Direct oral anticoagulant (DOACs) — Data of participants newly exposed to individual DOACs that is rivaroxaban, apixaban, dabigatran from 19-Oct-2010 to 31-Dec-2018 will be assessed. No study drug treatment will be administered as part of this observational study.
Drug: Warfarin — Data of participants newly exposed to warfarin from 19-Oct-2010 to 31-Dec-2018 will be assessed. No study drug treatment will be administered as part of this observational study.
  Groups: Comparator Group

SUMMARY:
The purpose of this study is assess the: (a) incidence of severe uterine bleeding (SUB) following exposure to individual direct oral anticoagulant (DOACs) (rivaroxaban, apixaban, dabigatran) and warfarin, (b) individual DOACs (rivaroxaban, apixaban, dabigatran) association with risk of SUB compared with warfarin, and (c) individual DOACs (rivaroxaban, apixaban, dabigatran) associated with risk of SUB compared with other individual DOACs - among women with prior diagnoses for DOAC and warfarin indications (non-valvular atrial fibrillation [NVAF], venous thromboembolism [VTE], total hip replacement [THR] or total knee replacement [TKR]).

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular atrial fibrillation (NVAF) diagnosis any time prior and no Venous thromboembolism (VTE) (Deep vein thrombosis [DVT] or Pulmonary embolism [PE]) in the past 183 days and no knee or hip replacement surgery in the past 35 days
* VTE (DVT or PE) in the past 183 days and no NVAF diagnosis any time prior and no knee or hip replacement surgery in the past 35 days
* Total hip replacement (THR) or Total knee replacement (TKR) in the past 35 days and no non-valvular atrial fibrillation any time prior and no venous thromboembolism (deep vein thrombosis of pulmonary embolism) in the past 183 days

Exclusion Criteria:

* Participants were excluded for edoxaban exposure, exposure to other exposures of interest (example: Direct oral anticoagulant [DOACs] for warfarin exposure cohort), hysterectomy, vaginal bleed, and medical, surgical, or transfusion management for vaginal bleeding any time prior to the index exposure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult women aged 18 years and older who are newly exposed to DOACs or warfarin with greater than or equal to (>=) 183 days of prior continuous database observation between 19-Oct-2010 and 31-Dec-2018 will be assessed for severe uterine bleeding.
Sampling Method: Probability Sample
Enrollment: 961985 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Severe Uterine Bleed | From 19-Oct-2010 to 31-Dec-2018
  Number of participants with severe uterine bleed during two time-at-risk periods (on-treatment and all observed time post-index) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen R&D, Titusville, New Jersey, United States

REFERENCES:
- [Derived] Weaver J, Shoaibi A, Truong HQ, Larbi L, Wu S, Wildgoose P, Rao G, Freedman A, Wang L, Yuan Z, Barnathan E. Comparative Risk Assessment of Severe Uterine Bleeding Following Exposure to Direct Oral Anticoagulants: A Network Study Across Four Observational Databases in the USA. Drug Saf. 2021 Apr;44(4):479-497. doi: 10.1007/s40264-021-01060-4. Epub 2021 Mar 2. PMID 33651368